CLINICAL TRIAL: NCT01079936
Title: Phase I/II Study Of The Combination Of Lenalidomide With High-Dose Melphalan For Autologous Transplant in Patients With Multiple Myeloma
Brief Title: Lenalidomide and High-Dose Melphalan
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0661; NCI-2011-00561 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Results first posted 2016-06-06 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-05

CONDITIONS: Myeloma; Stem Cell Transplantation
Keywords: Multiple Myeloma; Lenalidomide; Revlimid; Melphalan; Alkeran; Autologous stem cell transplantation; High-dose chemotherapy
MeSH Terms: conditions — Neoplasms, Plasma Cell; Multiple Myeloma | interventions — Lenalidomide; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide + High-Dose Melphalan (Experimental): Lenalidomide beginning dose level 25 mg by mouth (PO) on Days -8 to -2. High-Dose Melphalan dose level 100 mg/m2 by vein (IV) Days -3 and -2 over 30 minutes infusion. Stem cell infusion on Day 0.
  Interventions: Drug: Lenalidomide; Drug: Melphalan; Procedure: Stem Cell Infusion

INTERVENTIONS:
Drug: Lenalidomide — Beginning dose level 25 mg by mouth (PO) on Days -8 to -2
  Other Names: Revlimid; CC-5013
Drug: Melphalan — Dose level 100 mg/m2 by vein (IV) Days -3 and -2 over 30 minutes infusion
  Other Names: Alkeran
Procedure: Stem Cell Infusion — Stem cell infusion on Day 0.

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of the combination of Revlimid (lenalidomide) and high-dose Alkeran (melphalan) that can be given to patients with multiple myeloma who will receive an autologous stem cell transplantation. The safety of this combination therapy will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Melphalan is designed to damage the DNA (the genetic material of cells) of cells, which may cause cancer cells to die. High-dose melphalan is considered the standard of care for multiple myeloma.

Lenalidomide is designed to block a protein that plays a role in cell function and growth, which may cause cancer cells to die.

Study Dose Levels:

If you agree to take part in this study, you will be assigned to a dose level of lenalidomide based on when you join this study. Up to 4 dose levels of lenalidomide will be tested for safety. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen.

All participants will receive the same dose level of melphalan.

Once the highest tolerable dose of the combination of melphalan and lenalidomide is found, the next group of patients will be randomly assigned to 1 of 4 possible groups that will be determined by the computer, based on the safest and most effective dose level at that particular point.

Study Drug Administration:

You will take lenalidomide by mouth 1 time a day beginning 8 days before the stem cell transplant (Day -8). You will take the drug for 7 days (Days -8 through -2). You should take it with a few sips of water.

On Days -3 and -2, you will receive melphalan by vein over 30 minutes.

On Day 0, after you have received the chemotherapy study drugs, you will receive an infusion of stem cells, which were previously collected from you. This infusion of stem cells is given in an effort to help increase blood production and strengthen your immune system. You will receive antibiotics in an effort to decrease the likelihood that you will develop an infection.

Hospitalization following transplant usually lasts about 2-4 weeks, but may be longer. Some participants may be discharged earlier and followed in the outpatient clinic.

Study Visits:

About 1 month, 3 months, and 6 months after the transplant:

* You will have a physical exam and your medical history will be recorded.
* Blood (about 2 tablespoons) and urine will be collected for routine tests and to check the status of the disease.
* About 3 months after the transplant, you will have a bone marrow biopsy and aspiration to check the status of the disease. This will be repeated more often, if your doctor thinks it is needed.

About 1 year after the transplant:

* You will have a physical exam and your medical history will be recorded.
* Blood (about 2 tablespoons) and urine will be collected for routine tests.
* You will have a bone marrow biopsy and aspiration to check the status of the disease.
* You will have x-rays of your bones to check the status of the disease.

Length of Study:

Your participation in this study will be over after the 1 year transplant follow-up visit.

If intolerable side effects from the chemotherapy occur or there is sign of disease after the transplant, you will be taken off study. If you have intolerable side effects after you receive melphalan, then you will still have the transplant. However, if intolerable side effects develop before you take melphalan, you may be taken off study without having the transplant. If you are taken off study early, you still may need to return for routine post-transplant follow-up visits, if your transplant physician decides it is necessary.

It may be life-threatening to leave the study early during the conditioning regimen without following up with the stem cell transplant, because your blood cell counts may be dangerously low.

This is an investigational study. Lenalidomide and melphalan are commercially available and FDA approved for the treatment of myeloma. However, the use of lenalidomide with melphalan before an autologous stem cell transplant is investigational.

Up to 60 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with multiple myeloma with relapsed or progressive disease after achieving a partial or complete response to prior conventional therapy or autologous stem cell transplantation
2. Age 18 to 80 years
3. Performance score of at least 80% by Karnofsky or performance score of 0 or 1 (ECOG)
4. Left ventricular ejection fraction =/> 40%. No uncontrolled arrhythmias or symptomatic cardiac disease.
5. FEV1, FVC and DLCO=/> 40%. No symptomatic pulmonary disease.
6. Serum bilirubin <2 x upper limit of normal, SGPT <3x upper limit of normal. No evidence of chronic active hepatitis or cirrhosis. No pleural effusion or ascites > 1 L prior to drainage.
7. Creatinine Clearance =/> 50 ml/min
8. HIV negative
9. Negative beta HCG test in women with child bearing potential, defined as not post-menopausal for 24 months or no previous sterilization.
10. Patients or guardian able to sign informed consent.
11. All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
12. Females of childbearing potential (FCBP) must have a negative serum pregnancy test with a sensitivity of at least 50 mIU/mL within 10 -14 days prior to and again within 24 hours of prescribing lenalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 4 weeks before she starts taking lenalidomide.
13. Contd. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with females of child bearing potential even if they have had a successful vasectomy. See Appendix F: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods.

Exclusion Criteria:

1. Fertile men or women unwilling to use contraceptive techniques during and for 12 months following treatment.
2. Patients with uncontrolled hypertension (systolic > 140, diastolic >90 despite anti-hypertensive therapy.)
3. Patients with uncontrolled bacteria, viral or fungal infections (currently taking medication and progression of clinical symptoms).
4. Known hypersensitivity or desquamating rash to either thalidomide or lenalidomide.
5. Women who are pregnant (positive ß-HCG) or breastfeeding. (Lactating women must agree not to breast feed while taking lenalidomide and for 28 days after last dose of lenalidomide.)
6. New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmia's, or electrocardiographic evidence of acute ischemia, or a 2nd or 3rd degree AV block or new left bundle branch block on EKG.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muzaffar H. Qazilbash, MD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: March 01, 2010 to April 18, 2013. All recruitment done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Following Phase I portion of study, participants were assigned using adaptive randomization to 1 of 4 dose levels in Phase II. Out of 61 participants consented, 2 participants were ineligible for study due to first remission status and 2 participants did not receive stem cell transplant due to other issues and are not included in study demographic.
Groups:
- Phase I: Lenalidomide + High-Dose Melphalan: Lenalidomide beginning dose level 25 mg by mouth (PO) on Days -8 to -2. High-Dose Melphalan dose level 100 mg/m^2 by vein (IV) Days -3 and -2 over 30 minutes infusion. Stem cell infusion on Day 0.
- 25 Mg Lenalidomide: Lenalidomide dose level 25 mg by mouth (PO) on Days -8 to -2. High-Dose Melphalan dose level 100 mg/m^2 by vein (IV) Days -3 and -2 over 30 minutes infusion. Stem cell infusion on Day 0.
- 50 mg Lenalidomide: Lenalidomide dose level 50 mg by mouth (PO) on Days -8 to -2. High-Dose Melphalan dose level 100 mg/m^2 by vein (IV) Days -3 and -2 over 30 minutes infusion. Stem cell infusion on Day 0.
- 75 mg Lenalidomide: Lenalidomide dose level 75 mg by mouth (PO) on Days -8 to -2. High-Dose Melphalan dose level 100 mg/m^2 by vein (IV) Days -3 and -2 over 30 minutes infusion. Stem cell infusion on Day 0.
- 100 mg Lenalidomide: Lenalidomide dose level 100 mg by mouth (PO) on Days -8 to -2. High-Dose Melphalan dose level 100 mg/m^2 by vein (IV) Days -3 and -2 over 30 minutes infusion. Stem cell infusion on Day 0.
Period: Phase I: MTD
Arm/Group | Phase I: Lenalidomide + High-Dose Melphalan | 25 Mg Lenalidomide | 50 mg Lenalidomide | 75 mg Lenalidomide | 100 mg Lenalidomide
Started | 16 | 0 | 0 | 0 | 0
Completed | 12 (The 12 Phase I participants were randomized across 4 dose arms for Phase II.) | 0 | 0 | 0 | 0
Not Completed | 4 | 0 | 0 | 0 | 0
Not completed — First Remission Status | 2 | 0 | 0 | 0 | 0
Not completed — No Stem Cell Transplantation | 2 | 0 | 0 | 0 | 0
Period: Phase II
Arm/Group | Phase I: Lenalidomide + High-Dose Melphalan | 25 Mg Lenalidomide | 50 mg Lenalidomide | 75 mg Lenalidomide | 100 mg Lenalidomide
Started | 0 | 3 | 6 | 24 | 26
Completed | 0 | 3 | 5 | 24 | 25
Not Completed | 0 | 0 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0
Not completed — Insurance Issue | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Two participants were not eligible for study, and another two were eligible but did not receive required stem cell transplant therefore all appear in participation flow but two ineligible are not in baseline analysis population demographics.
Groups:
- Total: Total of all reporting groups
Arm/Group | 25 Mg Lenalidomide | 50 mg Lenalidomide | 75 mg Lenalidomide | 100 mg Lenalidomide | Total
Number analyzed (Participants) | 3 | 6 | 24 | 26 | 59
Age, Continuous [Median (Full Range); unit: years] | 59 [50 to 63] | 66 [53 to 70] | 55 [34 to 72] | 60 [52 to 71] | 59.5 [34 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 12 | 13 | 31
  Male | 1 | 2 | 12 | 13 | 28
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 24 | 26 | 59

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Lenalidomide
Description: There were 4 doses of lenalidomide in the dose escalation phase: 25 mg, 50 mg, 75 mg, and 100 mg. The first 12 patients were treated at these dose levels (3 patients per level) and safety assessed at each level. The MTD dose level was to be the level at which participants at each lenalidomide dose level had no dose limiting toxicity (DLT). DLT defined as as regimen-related death, graft failure, grade 3 or 4 atrial fibrillation, grade 4 deep venous thrombosis, or pulmonary embolism before day 30 after auto-HCT. Each participant received a fixed dose of Melphalan plus one of the four doses 25, 50, 75 or 100 mg of Lenalidomide orally for each of 7 days, -8 to -2 pre transplant.
Time Frame: Assessed at 21-28 Day Cycle
Population: Of the 16 participants in Phase I, two participants were not eligible for study due to first remission status, and two were eligible but did not receive stem cell transplant due to other issues.
Measure: Number; unit: mg/day
Arm/Group | Lenalidomide + High-Dose Melphalan
Number analyzed (Participants) | 12
mg/day | 100

2. Primary Outcome: Number of Participants With Response (CR at Day 90)
Description: Response is defined as the event that the participant is alive with complete response (CR) at day 90 (+/-30 days). CR defined as: A) Absence of monoclonal protein in urine and serum when analyzed by immunofixation electrophoresis. B) The bone marrow should be normal by morphological examination with <5% plasma cells. There should be < 1% aneuploid light chain restricted population by flow cytometry for DNA/cIg. C) While healing of bone lesions not required, no new lytic lesion should appear. Further compression fracture of spine will be not considered as progressive disease.
Time Frame: Day 90 after stem cell transplant
Measure: Number; unit: participants
Arm/Group | 25 Mg Lenalidomide | 50 mg Lenalidomide | 75 mg Lenalidomide | 100 mg Lenalidomide
Number analyzed (Participants) | 3 | 5 | 24 | 25
participants | 0 | 0 | 4 | 4

3. Primary Outcome: Number of Participants With Day 30 DLT (Overall Study, Phase I/Phase II)
Description: Dose limiting toxicity (DLT) was defined as regimen-related death, graft failure, grade 3 or 4 atrial fibrillation, grade 4 deep venous thrombosis, or pulmonary embolism before day 30 after auto-HCT.
Time Frame: Day 30 following transplant
Measure: Number; unit: participants
Arm/Group | 25 Mg Lenalidomide | 50 mg Lenalidomide | 75 mg Lenalidomide | 100 mg Lenalidomide
Number analyzed (Participants) | 3 | 5 | 24 | 25
participants | 0 | 0 | 2 | 0

4. Primary Outcome: Participants With Grade 3 =/> Adverse Events
Description: Number of participants experiencing adverse events above a Grade 3 according to the Common Terminology Criteria for Adverse Events (CTCAE) version 2.
Time Frame: Day 90 after stem cell transplant
Measure: Number; unit: participants
Arm/Group | 25 Mg Lenalidomide | 50 mg Lenalidomide | 75 mg Lenalidomide | 100 mg Lenalidomide
Number analyzed (Participants) | 3 | 5 | 24 | 25
participants | 3 | 5 | 15 | 17

ADVERSE EVENTS:
Time Frame: Adverse event collection from the start of preparative regiment up to Day 30 following stem cell transplant.
Arm/Group | 25 Mg Lenalidomide | 50 mg Lenalidomide | 75 mg Lenalidomide | 100 mg Lenalidomide
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/6 | 1/24 | 1/26
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 22/24 | 25/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 25 Mg Lenalidomide (N=3) | 50 mg Lenalidomide (N=6) | 75 mg Lenalidomide (N=24) | 100 mg Lenalidomide (N=26)
Blood Platelets (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 25 Mg Lenalidomide (N=3) | 50 mg Lenalidomide (N=6) | 75 mg Lenalidomide (N=24) | 100 mg Lenalidomide (N=26)
Change in Platelet levels (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
High blood pressure (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 9 (9) | 13 (13)
Herpetic lip leson (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
GU HEM (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Renal and urinary disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Hepatobiliary disorders (Renal and urinary disorders) | 0 (0) | 1 (1) | 4 (4) | 3 (3)
Infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 11 (11)
Other Neurologic Disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Other Skin Disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 4 (4)
Fever, Flu-like (General disorders) | 1 (1) | 0 (0) | 5 (5) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 6 (6) | 22 (22) | 21 (21)
GI DPH (Gastrointestinal disorders) | 2 (2) | 4 (4) | 10 (10) | 13 (13)
Infection, Neutropenic fever (Infections and infestations) | 2 (2) | 5 (5) | 9 (9) | 15 (15)
Nausea (Gastrointestinal disorders) | 3 (3) | 6 (6) | 22 (22) | 25 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes